CLINICAL TRIAL: NCT06477016
Title: A Randomized Pilot Study of the Efficacy of the OsciPulse System for the Reduction of Serum D-dimer
Brief Title: OsciPulse D-dimer Pilot Trial
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: OsciFlex LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: OSC-VTE-003
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group A-OsciPulse System: Patients admitted to the neuro intensive care unit or intermediate neurological care unit with a diagnosis of ischemic stroke randomly assigned to Group A.
  Interventions: Device: OsciPulse
- Group B- Standard Reference Therapy: Patients admitted to the neuro intensive care unit or intermediate neurological care unit with a diagnosis of ischemic stroke randomly assigned to Group B.
  Interventions: Device: Intermittent Pneumatic Compression

INTERVENTIONS:
Device: OsciPulse — Non-invasive device that provides rapid pulses of compression of the calves to modify venous blood flow patterns in immobilized persons.
  Groups: Group A-OsciPulse System
Device: Intermittent Pneumatic Compression — Non-invasive device that provides rapid pulses of compression of the calves to modify venous blood flow patterns in immobilized persons.
  Groups: Group B- Standard Reference Therapy

SUMMARY:
Pilot, randomized, non-blinded clinical trial to generate preliminary data to evaluate the impact of the OsciPulse system on serum d-dimer levels compared to standard of care intermittent compression therapy for DVT prophylaxis in patients admitted in the neuro ICU or intermediate neurological care unit with acute ischemic stroke.

DETAILED DESCRIPTION:
This is a single site, randomized open label two arm study. The patient population will be randomly divided into two arms, with one receiving the OsciPulse System and the other receiving standard intermittent compression therapy.

Both arms will have the therapy applied within 24 hours of admission and continue during their hospital stay until day 7 or discharge, whichever is shorter, unless clinically required to be removed. Daily d-dimer levels will be assessed until day 7 or discharge. If required beyond day 7, standard compression therapy will be provided. An interim analysis will be performed after 20 subjects are enrolled to evaluate the speed of enrollment and data variability and quality. If indicated, enrollment will be increased up to 40.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged ≥ 18 years old
2. Admitted to the Neuro Intensive Care Unit or Intermediate Neuro Care Unit with a diagnosis of ischemic stroke
3. Last known normal < 24 hours.
4. NIH stroke score ≥5
5. Weakness in at least one leg (≥ 1 point on the NIHSS lower extremity motor scores)
6. Prescribed mechanical therapy for DVT prophylaxis.

Exclusion Criteria:

1. Inability or contraindication to applying IPC to both legs such as:

* Evidence of acute bone fracture in lower extremities
* Acute burns in the lower extremities, lacerations, ulcers, active skin infection or dermatitis, in the lower extremities at the site of IPC placement
* Acute ischemia or severe peripheral vascular disease in the lower extremities as evidenced by cyanotic, cool, pulselessness.
* Amputated foot or leg on one or two sides
* Compartment syndrome (acute injury causing swelling and ischemic injury)
* Severe lower extremity edema (+4 edema as documented by clinical team)
* Acute deep vein thrombosis 2. Subjects who received thrombolytic therapy (e.g. Alteplase or Tenecteplase) for their stroke 3. Known pregnancy or within 6 weeks of postpartum period. 4. Limitation of life support, life expectancy < 7 days, or in hospice care 5. A head-unit is unavailable within 24 hours of last known normal. 6. At the discretion of the attending physician and / or clinical team, the subject's participation in the study is believed not to be in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects admitted to the Neuro ICU or Intermediate Neuro Care Unit with a diagnosis of acute stroke will be screened for enrollment.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in serum d-dimer levels. | 7 days
  Relative change in serum d-dimer levels for each subject from baseline to Day 7 or discharge

SECONDARY OUTCOMES:
Tolerability of the OsciPulse device in the stroke population | 7 days
  Tolerability defined as the number of patients who stop using the device prior to clinical recommendation and by quantitative scoring of subject experience questionnaires.
Safety of the OsciPulse device in the stroke population | 7 days
  Comparison of the rate of Adverse Events (AE) between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- HUP Neurology Dept. of Stroke and Neurocritical Care- University of Pennsylvania, Philadelphia, Pennsylvania, United States